CLINICAL TRIAL: NCT05271903
Title: A Simulation and Experiential Learning Intervention for Labor and Delivery Providers to Address HIV Stigma During Childbirth in Tanzania
Brief Title: Simulation Training for Labor and Delivery Providers to Address HIV Stigma During Childbirth in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Melissa Watt, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R21TW012001-01 (NIH); R21TW012001 (NIH)
Record Dates: First submitted 2022-02-16; First posted 2022-03-09 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hiv; Stigmatization; Pregnancy Related
Keywords: HIV; stigma; childbirth; simulation training
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Stereotyping; Social Stigma

STUDY DESIGN:
Intervention Model Description: MAMA intervention: a simulation training for labor and delivery providers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The MAMA intervention, which is a simulation training intervention for labor and delivery prviders.
  Interventions: Behavioral: MAMA Intervention

INTERVENTIONS:
Behavioral: MAMA Intervention — The MAMA intervention will be based on PRONTO International's simulation training program to improve obstetric care delivery. The PRONTO curriculum is based on simulation and debrief of clinical scenarios, case-based learning, skills stations, and interactive teamwork and communication activities. Through the training, providers review and learn clinical skills related to obstetric care and emergencies, while reflecting on and practicing principles of respectful maternity care. The simulation exercises give providers and opportunity to "act" as the patient and develop empathy for the patient experience, and debriefing after simulation includes a reflection and discussion about RMC principles. The training will be two full days, followed by a refresher training in the clinical setting after one month.

SUMMARY:
This study will work in Tanzania to develop and pilot test a simulation and experiential learning intervention for labor and delivery providers, in order to address HIV stigma during childbirth. The primary endpoint will be patient-rated changes in respectful maternity care, comparing women who deliver in the pre-intervention time period and women who deliver in the post-intervention period.

DETAILED DESCRIPTION:
The study will pilot test the MAMA intervention in six clinics in the Kilimanjaro Region. 60 L&D providers will be enrolled across the sites. Patient level outcomes will be assessed using an interrupted time series design. Approximately 206 participants will be enrolled (103 in the pre-intervention period and 103 in the post-intervention period). The primary outcome will be patients' reported experiences of respectful maternity care (RMC). Secondary outcomes will be internalized HIV stigma, trust in health care, birth outcomes, HIV care engagements at 3 months, anticipated HIV stigma, and attitudes to long-term antiretroviral therapy. Our enrollment targets (103 per condition) will allow for detection of a medium effect of 0.4 in the change of RMC overall scores with 80% power and α=0.05. Pre- and post- surveys will be conducted for providers enrolled in the intervention, assessing outcomes related to practices of RMC, stigma toward WLHIV, self efficacy and clinical knowledge.

ELIGIBILITY:
Inclusion Criteria:

Labor and delivery providers who are:

* Over age 18
* Employed by a study clinic
* Work in the labor and delivery ward

Exclusion Criteria:

* Has not provided clinical care in the labor and delivery ward in past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: No
The data from the formative and pilot trial work in this R21 will be freely shared within the constraints required for the protection of confidentiality for study subjects. With a data transfer agreement from out Institutional Review Board, we are willing to share raw data with researchers and program leaders from other institutions.

REFERENCES:
- [Derived] Hanson OR, Weglarz AJ, Barabara ML, Cohen SR, Minja LM, Mlay PS, Stephens MJ, Olomi GA, Mlay J, Mmbaga BT, Watt MH. HIV-related Shame among Women Giving Birth in Tanzania: A Mixed Methods Study. AIDS Behav. 2024 Jul;28(7):2276-2285. doi: 10.1007/s10461-024-04322-1. Epub 2024 Mar 25. PMID 38526642
- [Derived] Watt MH, Minja LM, Barabara M, Mlay P, Stephens MJ, Olomi G, Mlay J, Marchand V, Mmbaga BT, Hanson OR, Cohen SR. A simulation and experiential learning intervention for labor and delivery providers to address HIV stigma during childbirth in Tanzania: study protocol for the evaluation of the MAMA intervention. BMC Pregnancy Childbirth. 2023 Mar 16;23(1):181. doi: 10.1186/s12884-023-05482-z. PMID 36927460
- [Derived] Watt MH, Cohen SR, Minja LM, Barabara M, Mlay P, Stephens MJ, Olomi G, Mlay J, Marchand V, Mmbaga BT. A simulation and experiential learning intervention for labor and delivery providers to address HIV stigma during childbirth in Tanzania: Study protocol for the evaluation of the MAMA intervention. Res Sq [Preprint]. 2023 Jan 30:rs.3.rs-2285235. doi: 10.21203/rs.3.rs-2285235/v1. PMID 36778232

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this pilot trial, the primary outcome measure (change in respectful maternity care score) was assessed with the health care providers (n=60) who were enrolled and exposed to the MAMA training intervention.
Groups:
- MAMA Training: 2.5 day health care provider simulation training for respectful and non-stigmatizing labor and delivery care for people living with HIV.
Period: Overall Study
Arm/Group | MAMA Training
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 60
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Respectful Maternity Care
Description: Practices of respectful maternity care were assessed using the measure "Person-centered maternity care" that Afulani et al validated in Kenya and Ghana. The scale includes nine questions that asked how often they had used person-centered practices in the past month. Items had four response options (never to always) and were summed. Scale has a possible range of 0 to 27, with higher values reflecting better outcomes (i.e., more respectful care).
Time Frame: 3 months
Population: Includes only the health care providers (n=60) who received the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MAMA Training
Number analyzed (Participants) | 60
score on a scale | 21.8 (3.1)

ADVERSE EVENTS:
Time Frame: Intervenmtion period (2.5 days)
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT05271903/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT05271903/SAP_001.pdf